CLINICAL TRIAL: NCT03372785
Title: The Success of Opening Concurrent Chronic Total Occlusion leSion to Improve Cardiac Function Trial in Patients With Multi-vessel Disease (SOS-moral): Study Protocol of a Prospective Multicenter Study
Brief Title: The Success of Opening Concurrent CTO leSion to Improve Cardiac Function Trial in Patients With Multi-vessel Disease
Acronym: SOS-moral
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Beijing Anzhen Hospital (Other)
Collaborators: The First Affiliated Hospital of Dalian Medical University (Other); Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Xiantao Song, MD, Professor, Beijing Anzhen Hospital
Other Study IDs: SOS-moral
Record Dates: First submitted 2017-12-10; First posted 2017-12-14 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Chronic Total Occlusion of Coronary Artery; Percutaneous Coronary Intervention; Coronary Artery Disease; Viable Myocardium
Keywords: Chronic total coronary artery occlusion; multi-vessel coronary artery disease; Percutaneous coronary intervention; coronary artery disease; cardiac function
MeSH Terms: conditions — Coronary Artery Disease | interventions — Aspirin; Metoprolol; Atorvastatin; Rosuvastatin Calcium; Clopidogrel; Ticagrelor; Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Complete revascularization group: Complete Revascularization of CTO and non-CTO lesions
  Interventions: Drug: aspirin, betaloc, atorvastatin, rosuvastatin, clopidogrel, ticagrelor; Device: coronary wires. stents or coronary balloons
- Non-CTO revascularization group: Non-CTO vessel revascularization
  Interventions: Drug: aspirin, betaloc, atorvastatin, rosuvastatin, clopidogrel, ticagrelor; Device: coronary wires. stents or coronary balloons

INTERVENTIONS:
Drug: aspirin, betaloc, atorvastatin, rosuvastatin, clopidogrel, ticagrelor — Optimal medical therapy includes dual antiplatelet therapy and statins (aspirin, clopidogrel, ticagrelor, atorvastatin, rosuvastatin, betaloc). And optimal medical therapy should include adequate ventricular rate-limiting medication (i.e. Beta-blocker or rate-limiting calcium antagonist) where appropriate. Anti-anginal therapy should be used if the patients have symptom.
  Other Names: Optimal medical therapy
Device: coronary wires. stents or coronary balloons — all species of drug-eluting stent ((such as Xience, Endeavor, Resolute) implantation or balloon expansion (POBA)
  Other Names: percutaneous coronary intervention

SUMMARY:
The purpose of this study is to investigate the effect of percutaneous coronary intervention (PCI) on cardiac function in multi-vessel disease patients with concurrent chronic total occlusion (CTO) lesion.

DETAILED DESCRIPTION:
Recruited CTO patients will be devided into two groups: those undergoing PCI of only the non-CTO artery (non-CTO PCI group), and those undergoing PCI of the non-CTO artery concurrently with the CTO artery (CTO-PCI group). The primary outcome assessed will be the change in cardiac function evaluated via CMR at a 12-month of follow-up appointment, which will be compared to a baseline measurement. Secondary outcomes include occurrence of major cardiac events, CMR-assessed myocardial viability in the CTO-supplied territory, and quality of life assessed by Seattle angina questionnaire, Patient Health Questionnaire 9 and Generalized Anxiety Disorder Scale-7 after 12-month follow-up.

ELIGIBILITY:
Inclusion criteria:

Patients should be 18-80 years old; be diagnosed with single CTO concurrent with MVD detected using coronary angiography (at least one other major vessel should have exhibited no less than 75% stenosis); present with an LVEF above 35% determined using transthoracic echocardiography; present with CTO located in an epicardial coronary artery with a reference diameter of ≥ 2.5 mm; and comply all the evaluations and follow-up protocols.

Exclusion criteria:

Patients will be excluded if they have suffered from acute myocardial infarction within the previous 3 months; a lesion located in the left main artery (stenosis ≥50%); rheumatic valvular disease; severe arrhythmia; a history of revascularization within the non-CTO artery; multiple vessels with CTO (more than one CTO artery); lesions unsuitable for PCI; severely abnormal hematopoietic systems, such as platelet counts <100 x 109/L or > 700 x 109/L and white blood cell counts < 3 x 109/L; with active bleeding or bleeding tendencies (active ulcers, short-term ischemic stroke, history of hemorrhagic stroke, intracranial space occupying lesions, recent craniocerebral trauma, and other bleeding or bleeding tendency); severe coexisting conditions, including severe renal function dysfunction [Glomerular filtration rate (GFR) less than 60 ml/min • 1.73 m2), severe hepatic dysfunction [glutamic-pyruvic transaminase (ALT) or glutamic-oxal acetic transaminase (ALT) elevated more than three times that of the upper limit of the normal reference], severe heart failure (NYHA classification III-IV), acute infectious diseases and immune disorders; tumors; surgery within 3 months; a life expectancy less than 12 months; pregnancy or planning to become pregnant; history of allergy or adverse reactions to aspirin, clopidogrel, ticagrelor, stains, contrast material, anticoagulant, or stents. Patients will also be excluded if they cannot tolerate dual antiplatelet treatment (DAPT); are unable to communicate due to cognitive impairment, auditory, or visual impairment; are participating in another trial for medication or an apparatus and in which the main endpoint has not been reached, or plan to participate in a clinical trial within 12 months of the intervention.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients should be 18-80 years old; be diagnosed with single CTO concurrent with MVD detected using coronary angiography (at least one other major vessel should have exhibited no less than 75% stenosis); present with an LVEF above 35% determined using transthoracic echocardiography; present with CTO located in an epicardial coronary artery with a reference diameter of ≥ 2.5 mm; and comply all the evaluations and follow-up protocols
Sampling Method: Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2018-04-10 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Changes of left ventricular ejection fraction (LVEF) | 12 months
  Changes of LVEF, LVEDV, and LVESV assessed with the use of cardiac MRI.

SECONDARY OUTCOMES:
Major adverse cardiac events | 1, 6, and 12 months post-PCI
  all-cause mortality, cardiac death, a first or recurrent, non-fatal, acute myocardial infarction, target lesion revascularization (PCI or CABG), stroke, heart failure and cardiac rehospitalization
Myocardial viability | 12 months post-PCI
  myocardial viability in the territory supplied by the CTO artery
Quality of life changes | 1, 6, and 12-month follow-up
  Seattle Angina Questionnaire, Patient Health Questionnaire 9 and Generalized Anxiety Disorder Scale-7
Contrast used | during the procedure
  contrast used
Total cost of medical care | from the day of enrollment (first hospitalization) to the last follow-up (rehospitalization)
  total cost of medical care covering optimal medicine therapy and the equipment for coronary artery disease therapy from the day of enrollment (first hospitalization) to the last follow-up (rehospitalization)

OTHER OUTCOMES:
Safety endpoints | perioperative period
  The safety of the perioperative period, including acute coronary artery occlusion, acute vascular perforation, acute stent thrombosis, acute myocardial infarction, and cardiac death

CONTACTS AND LOCATIONS:
Overall Officials: Xiantao Song, MD, Principal Investigator — Beijing Anzhen Hospital
Locations (1):
- Department of Cardiology, Beijing Anzhen Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided